CLINICAL TRIAL: NCT00833846
Title: Pilot Study of Mitochondrial Biology in Human Platelets
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090068; 09-H-0068
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-10-24

CONDITIONS: Insulin Resistance; Diabetes
Keywords: Mitochondria in Platelets; Mitochondria in Diabetes; Insulin Resistance and Mitochondria; Diabetes; Insulin Resistance
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Type II diabetes mellitus is rapidly becoming a global pandemic with a deleterious impact on cardiovascular morbidity and mortality. Understanding its pathophysiology is important for the development of future therapeutic interventions. Emerging evidence suggests interplay between mitochondrial dysfunction and the development of insulin resistance. Interestingly, mitochondrial dysfunction in skeletal muscle and adipose tissue are early events in the development of type II diabetes mellitus and are proposed to play a role in exacerbating insulin resistance. Although it has been demonstrated that skeletal muscle of insulin-resistant individuals has reduced mitochondria and mitochondrial dysfunction, whether this disruption of mitochondrial function is more widespread has not been explored. We hypothesize that this disruption of mitochondrial function is more systemic and thereby may contribute to the development of peripheral insulin resistance and possibly promote the myriad of complications associated with diabetes.

To test these assumptions, we propose an initial proof of concept study to evaluate mitochondrial biology in human platelets in normal volunteers, pre-diabetic and diabetic subjects to assess whether mitochondrial disruption/dysfunction evolves with the progression to type II diabetes. In parallel, proteomic analysis will be performed to evaluate whether the development of insulin resistance and diabetes confers a specific modulation in the biological signature of human platelets with disease progression. To delineate these concepts, we will evaluate study subject's glucose tolerance and insulin sensitivity and draw blood in parallel to study their platelets. Biological readouts will include: 1) the quantification of the mitochondrial proteome and electron transfer chain content; 2) the evaluation of platelet mitochondrial respiratory function and 3) to determine the mitochondrial reactive oxygen species capacity and defenses. If this hypothesis is validated, this study will show that the mitochondrial disruption/dysfunction is a more generalized finding in type II diabetes. Additionally, it would propose the use of platelets as potential biomarkers for early detection of mitochondrial function and assessment of disease. Finally, this would establish a peripheral blood readout of the modification of mitochondrial function as a novel approach to monitor the prevention and/or reversal of insulin resistance and diabetes in response to therapeutic strategies.

DETAILED DESCRIPTION:
Type II diabetes mellitus is rapidly becoming a global pandemic with a deleterious impact on cardiovascular morbidity and mortality. Understanding its pathophysiology is important for the development of future therapeutic interventions. Emerging evidence suggests interplay between mitochondrial dysfunction and the development of insulin resistance. Interestingly, mitochondrial dysfunction in skeletal muscle and adipose tissue are early events in the development of type II diabetes mellitus and are proposed to play a role in exacerbating insulin resistance. Although it has been demonstrated that skeletal muscle of insulin-resistant individuals has reduced mitochondria and mitochondrial dysfunction, whether this disruption of mitochondrial function is more widespread has not been explored. We hypothesize that this disruption of mitochondrial function is more systemic and thereby may contribute to the development of peripheral insulin resistance and possibly promote the myriad of complications associated with diabetes.

To test these assumptions, we propose an initial proof of concept study to evaluate mitochondrial biology in human platelets in normal volunteers, pre-diabetic and diabetic subjects to assess whether mitochondrial disruption/dysfunction evolves with the progression to type II diabetes. In parallel, proteomic analysis will be performed to evaluate whether the development of insulin resistance and diabetes confers a specific modulation in the biological signature of human platelets with disease progression. To delineate these concepts, we will evaluate study subject's glucose tolerance and insulin sensitivity and draw blood in parallel to study their platelets. Biological readouts will include: 1) the quantification of the mitochondrial proteome and electron transfer chain content; 2) the evaluation of platelet mitochondrial respiratory function and 3) to determine the mitochondrial reactive oxygen species capacity and defenses. If this hypothesis is validated, this study will show that the mitochondrial disruption/dysfunction is a more generalized finding in type II diabetes. Additionally, it would propose the use of platelets as potential biomarkers for early detection of mitochondrial function and assessment of disease. Finally, this would establish a peripheral blood readout of the modification of mitochondrial function as a novel approach to monitor the prevention and/or reversal of insulin resistance and diabetes in response to therapeutic strategies.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Inclusion Criteria (young control group):

1. Adults older than 21 years and less than 40 years.
2. Insulin sensitivity with a fasting glucose less than 100 mg/dl and a 2-hour post oral glucose tolerance test blood glucose less than 140 mg/dl.
3. Subject understands protocol and provides written, informed consent.

Inclusion Criteria (young insulin-resistant group):

1. Adults older than 21 years and less than 40 years.
2. Insulin resistance as defined by a fasting blood sugar of greater than or equal to 100mg/dl but less than 125 mg/dl and/or a 2-hour post oral glucose tolerance test blood glucose greater than 140 mg/dl and less than 200 mg/dl.
3. Subject understands protocol and provides written, informed consent.

Inclusion Criteria (middle age control group):

1. Adults greater than or equal to 40 years and less than or equal to 60 years.
2. Insulin sensitivity with a fasting blood glucose less than 100 mg/dl and a 2-hour post oral glucose tolerance test blood glucose less than 140 mg/dl.
3. Subject understands protocol and provides written, informed consent.

Inclusion Criteria (middle age insulin-resistant group):

1. Adults greater than or equal to 40 years and less than or equal to 60 years.
2. Insulin resistance as defined by a fasting blood sugar of greater than or equal to 100mg/dl but less than 125 mg/dl and/or a 2-hour post oral glucose tolerance test blood glucose greater than 140 mg/dl and less than 200 mg/dl.
3. Subject understands protocol and provides written, informed consent.

Inclusion Criteria (middle age type II diabetes group):

1. Adults greater than or equal to 40 years and less than or equal to 60 years.
2. Type II diabetes as defined by a fasting blood sugar of greater than 125 mg/dl and/or a 2-hour post oral glucose tolerance test blood glucose greater than 200 mg/dl if untreated and/or if subjects are on oral hypoglycemic agent therapy where the HbA1c is greater than 6.7 percent.
3. Subject understands protocol and provides written, informed consent.

Exclusion Criteria (all study subjects) :

1. Uncontrolled hypertension, heart failure, unstable coronary artery disease or symptomatic peripheral arterial disease requiring changes in medication or medical intervention in the preceding 3 months.
2. Insulin-dependant diabetes mellitus or current use of thiazolidinediones.
3. Women of childbearing age unless recent pregnancy test is negative and are not breast feeding.
4. Serum creatinine greater than 2.5 mg/dl.
5. Liver transaminase levels greater than 2.5 times upper limit of normal.
6. History of cancer treated with chemotherapy or irradiation in the last 5 years.
7. Active inflammatory disease, or infection, or abnormal white blood cell differential.
8. Enrollment in any drug studies within the last 30 days.
9. BMI greater than 35 for the middle age groups and greater than 30 for the younger subjects.
10. Age greater than 60 years.
11. Another member of a potential study subject's immediate family has been recruited/participated in this study.
12. The use of anticoagulation therapy, thiazide diuretics, corticosteroids, or some psychiatric drugs that cannot be stopped for medical reasons for a few days for study participation.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-01-27; Study Completion 2011-10-24

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Barr EL, Zimmet PZ, Welborn TA, Jolley D, Magliano DJ, Dunstan DW, Cameron AJ, Dwyer T, Taylor HR, Tonkin AM, Wong TY, McNeil J, Shaw JE. Risk of cardiovascular and all-cause mortality in individuals with diabetes mellitus, impaired fasting glucose, and impaired glucose tolerance: the Australian Diabetes, Obesity, and Lifestyle Study (AusDiab). Circulation. 2007 Jul 10;116(2):151-7. doi: 10.1161/CIRCULATIONAHA.106.685628. Epub 2007 Jun 18. PMID 17576864
- [Background] Morino K, Petersen KF, Shulman GI. Molecular mechanisms of insulin resistance in humans and their potential links with mitochondrial dysfunction. Diabetes. 2006 Dec;55 Suppl 2(Suppl 2):S9-S15. doi: 10.2337/db06-S002. PMID 17130651
- [Background] Lowell BB, Shulman GI. Mitochondrial dysfunction and type 2 diabetes. Science. 2005 Jan 21;307(5708):384-7. doi: 10.1126/science.1104343. PMID 15662004